CLINICAL TRIAL: NCT05207267
Title: Safety of Driving Pressure-guided Tidal Volume Setting in ARDS Patients-From the Perspective of EIT
Brief Title: Driving Pressure Guided VT in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ling-driving pressure
Record Dates: First submitted 2021-08-20; First posted 2022-01-26 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: ARDS
Keywords: ARDS; ventilation and perfusion matching; ventilation inhomogeneity
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- testing arm (Experimental): ventilated with different VT using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany)
  Interventions: Device: driving pressure guided tidal volume

INTERVENTIONS:
Device: driving pressure guided tidal volume — Volume control mode without spontaneous breathing, PEEP will be set according to best respiratory compliance method, and tidal volume (VT) will be set to reach three levels of driving pressure (High 14-15cmH2O, moderate 10-11 cmH2O, and low 7-8 cmH2O). Each level of VT was maintained 10 minutes in supine and/or prone position.

SUMMARY:
A prospective physiologic study, in participants with COVID-19 related or non-COVID-19 related acute respiratory distress syndrome (ARDS) requiring mechanical ventilation less than 48 hours. The investigators assessed the effect of different tidal volume guided by different levels of driving pressure on ventilation inhomogeneity and ventilation/perfusion mismatch by electrical impedance tomography (EIT) in supine and/or prone position.

DETAILED DESCRIPTION:
Once enrolled, an EIT dedicated belt containing 16 electrodes was placed around the participant's chest at the fifth or sixth intercostal space and connected it to an EIT monitor (PulmoVista 500; Dräger Medical GmbH, Lübeck, Germany).

Data were collected in the enrolled day (Day 1),Day 3 and Day 7 including demographic and anthropometric data, a baseline arterial blood gas measurement, and ventilation parameters including type of supplemental oxygen, respiratory rate, fractional concentration of oxygen in inspired air (FiO2).

Volume control mode without spontaneous breathing, PEEP will be set according to best respiratory compliance method, and tidal volume (VT) will be set to reach three levels of driving pressure (High 14-15cmH2O, moderate 10-11 cmH2O, and low 7-8 cmH2O). Each level of VT was maintained 10 minutes in supine and/or prone position. In the last minutes of each phase，the participants received instructions of end expiratory occlusion lasting at least 10 seconds and, 1 seconds after the start, a bolus of 10 mL of 10% NaCl solution was injected via the central venous catheter. Clinical data and outcome will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years old
2. admitted to intensive care unit with a moderate to severe ARDS
3. invasive mechanical ventilation

Exclusion Criteria:

1. contraindications for prone position ventilation
2. Past chronic respiratory diseases (long-term family oxygen therapy for chronic respiratory diseases such as pulmonary fibrosis or COPD)
3. New York Heart Association class above II
4. gave written or witnessed verbal informed consent.
5. Contraindications to the use of EIT (e.g., presence of pacemaker or chest surgical wounds dressing) or prone position (as decided by the attending physician)
6. Impending ECMO (on the basis of clinical judgment, including clinical and physiological parameters).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
regional compliance using EIT | Day 1
  regional compliance using EIT
regional ventilation | Day 1
  regional ventilation using EIT
regional perfusion | Day 1
  regional perfusion using EIT
Region-ventilation-delay | Day 1
  Region-ventilation-delay using EIT
driving pressure | Day 3
  measurement as one index of respiratory compliance
the number of regional lung ventilation | Day 3
  regional ventilation measuring by EIT
the number of regional lung perfusion | Day 3
  regional perfusion measuring by EIT
the number of region-ventilation-delay (RVD) | Day 3
  the RVD measuring by EIT

SECONDARY OUTCOMES:
Value of ventilation-perfusion (V/Q) mismatch | Day 1
  V/Q mismatch was quantified as the percentage of pixels that were classified as ventilated but not perfused (dead space fraction) plus the percentage of those perfused but not ventilated (shunt fraction).
Value of ventilation-perfusion (V/Q) mismatch | Day 3
  V/Q mismatch was quantified as the percentage of pixels that were classified as ventilated
Value of ventilation-perfusion (V/Q) mismatch | Day 7
  V/Q mismatch was quantified as the percentage of pixels that were classified as ventilated
The Global Inhomogeneity (GI) index | Day 1
  higher values indicating less homogenous ventilation
The Global Inhomogeneity (GI) index | Day 3
  higher values indicating less homogenous ventilation
The Global Inhomogeneity (GI) index | Day 7
  higher values indicating less homogenous ventilation
Blood gas | Day 1
  PaO2
Ventilation free day | Day 28
  ventilation free day in day 28
28 day mortality | Day 28
  death in day 28

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, Study Director — Zhongda Hospital, School of Medicine, Southeast Univerty
Locations (1):
- Ling Liu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
by email
Supporting Information: Study Protocol, SAP, CSR
Time Frame: with in two years after publication
Access Criteria: other researchers

REFERENCES:
- [Derived] Yuan X, Zhao Z, Chao Y, Chen D, Chen H, Zhang R, Liu S, Xie J, Yang Y, Qiu H, Heunks L, Liu L. Effects of early versus delayed application of prone position on ventilation-perfusion mismatch in patients with acute respiratory distress syndrome: a prospective observational study. Crit Care. 2023 Nov 27;27(1):462. doi: 10.1186/s13054-023-04749-3. PMID 38012731